CLINICAL TRIAL: NCT01091220
Title: A Randomized, Single-center, Double-blind, Placebo-controlled Study to Explore the Effect of a Single Dose of Certolizumab Pegol 400 mg on Semen Quality in Healthy Male Volunteers
Brief Title: Evaluation of the Effects of Certolizumab Pegol on Semen Quality in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CR0001; 2009-015216-17 (EudraCT Number)
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-03

CONDITIONS: Sperm Quality
Keywords: certolizumab pegol; Cimzia®; healthy male volunteers; sperm
MeSH Terms: interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 0.9% saline
  Interventions: Biological: Placebo
- Certolizumab pegol (Experimental): Certolizumab pegol 400 mg
  Interventions: Biological: Certolizumab pegol

INTERVENTIONS:
Biological: Certolizumab pegol — 400 mg certolizumab pegol in 2 x 200 mg/mL, prefilled syringes, administered once, subcutaneously
  Other Names: Cimzia®
  Arms: Certolizumab pegol
Biological: Placebo — 2 x prefilled syringes containing 0.9% saline, administered once, subcutaneously
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of certolizumab pegol (CZP) on the quality of sperm obtained from healthy male volunteers.

DETAILED DESCRIPTION:
CZP is a PEGylated humanized Fab' fragment with specificity for human tumor necrosis factor alpha (TNFα). Evidence suggests that modulation of TNFα signaling may affect male spermatogenesis. Therefore, this study will compare semen quality parameters before and after a single 400 mg dose of CZP, or matched placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers with normal baseline semen quality parameters

Exclusion Criteria:

* Previous participation in studies involving TNF inhibitors
* Prior treatment with biologic response modifiers within 5 half-lives
* History of trauma or surgery to the pelvis/genital area
* Tests positive for tuberculosis, HIV, Hepatitis B or C

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Total sperm motility (%) | baseline to 99 days
Sperm morphology (%) | Baseline to 99 days

SECONDARY OUTCOMES:
Progressive motility (%) | Baseline to 99 days
Non-progressive motility (%) | Baseline to 99 days
Sperm vitality (%) | Baseline to 99 days
Semen volume (mL) | Baseline to 99 days
Sperm count (millions) | Baseline to 99 days
Sperm concentration (millions/mL) | Baseline to 99 days

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Liège, Belgium